CLINICAL TRIAL: NCT06120192
Title: Examining the Effect of Piano Playing Training on Fine Motor Skills in Parkinson's Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of staff
Sponsor: Tel Aviv University (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Jason Friedman, Associate Professor, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8407-21-SMC
Record Dates: First submitted 2023-10-26; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: music; piano; dexterity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Open label feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research group (Experimental): Receives the full piano training
  Interventions: Behavioral: Piano

INTERVENTIONS:
Behavioral: Piano — Receives the piano training

SUMMARY:
Piano playing may provide an engaging and accessible setting for finger and wrist movement training. Moreover, it has been found effective for improving manual dexterity and upper-limb function in other neurologic disorders, such as stroke and additionally beneficial for cognitive and psychosocial support in Parkinson's disease. However, no study has examined the effect of piano playing on dexterity in Parkinson's disease. The aim of this study is to test the efficacy of a novel piano-based training program on fine motor function in patients with PD. Participants with Parkinson's disease will take part in an individually tailored 6-week piano training program, combining weekly supervised training sessions (6x60 min altogether), with three independent at-home weekly 30 minutes practice sessions (18x30 altogether). Participants will receive a piano MIDI keyboard for home use during the study.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease patients
* Hoehn and Yahr stages I to III
* Self-reports of some dexterity difficulties

Exclusion Criteria:

* Participation in an ongoing clinical study or clinical study within 30 days prior to this study
* Atypical parkinsonian syndrome or secondary parkinsonism (e.g., due to drugs, metabolic neurogenetic disorders, encephalitis, cerebrovascular disease, or other degenerative disease), or other neurologic conditions influencing upper limb movement
* Significant psychiatric symptoms or history
* Significant or recent experience in piano playing (participants who are proficient piano players, or had studied piano for more than 3 years in the past, or for shorter periods in the last 5 years)
* Other significant fine motor skills (e.g., high proficiency in playing another musical instrument, video games, etc.)
* Mini Mental status examination (MMSE) score below 25
* Significant sensory deficits, e.g., hearing or sight impairment
* Unstable medical disorder
* Significant postural or action tremor, moderate dyskinesia

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Box and block test | First meeting, last meeting (after 6 weeks)
  Number of blocks that can be moved over a barrier using the hand / arm in one minute
9 Hole peg test | First meeting, last meeting (after 6 weeks)
  Time taken to insert 9 pegs into holes and then remove them
Synergy index | First meeting, last meeting (after 6 weeks)
  Calculated from a force ramp production task using the fingers with force sensors
Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) motor parts II (patient questionnaire) - parts 2.4 to 2.7 and III (motor examination) - parts 3.3 and 3.4 | First meeting, last meeting (after 6 weeks)
  Standard questionnaire used in Parkinson's disease. Higher scores indicate more impairment. Maximum score for each part is 4, so overall for the 6 parts the maximum score is 24.

SECONDARY OUTCOMES:
Quantitative Digitography - Average strike duration | First meeting, last meeting (after 6 weeks)
  Measure of speed and variability of key presses on a piano - mean of the time the key is pressed
Quantitative Digitography - Coefficient of variation strike duration | First meeting, last meeting (after 6 weeks)
  Measure of speed and variability of key presses on a piano - coefficient of variation of the time the key is pressed
Quantitative Digitography - Average interval between strikes (in seconds) | First meeting, last meeting (after 6 weeks)
  Measure of speed and variability of key presses on a piano - average time between subsequent key presses
Quantitative Digitography - Coefficient of variation of interval between strikes | First meeting, last meeting (after 6 weeks)
  Measure of speed and variability of key presses on a piano - coefficient of variation of the time between subsequent key presses
Quantitative assessment of piano performance progress | First meeting, last meeting (after 6 weeks)
  Measurement of improvement in playing the piano - the teacher (rater) will give a score (between 0 and 5) for the level of piano playing of the participant, where 0 is no ability to play and 5 is the ability to play the pieces from the workbook (a beginner's level piano book) perfectly.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
Anonymous raw data from the tests will be made available on figshare
Supporting Information: ICF
Time Frame: Upon publication
Access Criteria: Open to all

REFERENCES:
- Available data/document: Informed Consent Form: 10.6084/m9.figshare.23994768 — https://doi.org/10.6084/m9.figshare.23994768
- Available data/document: Individual Participant Data Set: 10.6084/m9.figshare.23994768 — https://doi.org/10.6084/m9.figshare.23994768